CLINICAL TRIAL: NCT03102866
Title: Can Aerobic and Strength Training Exercise Initiated During and Continued After Radiation Therapy for Breast Cancer Improve Fitness and Arm Health 1 Year Later?
Brief Title: Aerobic and Strength Training Exercise in Improving Fitness and Arm Health During and After Radiation Therapy in Patients With Stage II-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sasha Beyer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-16125; NCI-2017-00318 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-03-20; First posted 2017-04-06 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients receive usual care for 6 weeks during radiation therapy and for 12 weeks after completion of radiation therapy.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (aerobic and strength training exercise) (Experimental): Patients undergo a supervised aerobic and strength training exercise session over 40-60 minutes 3 times weekly for 6 weeks during radiation therapy and for 12 weeks after completion of radiation therapy.
  Interventions: Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm I (usual care)
Behavioral: Exercise Intervention — Undergo aerobic and strength training exercise
  Arms: Arm II (aerobic and strength training exercise)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot phase I/II trial studies how well aerobic and strength training exercise works in improving fitness and arm health during and after radiation therapy consisting of regional nodal radiation in patients with stage II-III breast cancer. Aerobic and strength training exercise training during and after radiation therapy may reduce treatment related toxicities and improve adherence to exercise long term in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of conducting an exercise program during and after radiation therapy and to determine what percent of patients will complete the exercise program. (Pilot) II. To determine the percent increase in fitness as measured by the 6 minute walk test in women receiving radiation therapy for breast cancer randomized to an exercise program at 1 year. (Phase II)

SECONDARY OBJECTIVES:

I. Percent adherence to exercise at 1 year as measured by the International Physical Activity Questionnaire and exercise logs.

II. Subjective arm health at 1 year as measured by Functional Assessment of Cancer Therapy Questionnaire for Breast Cancer version 4 (FACT-B+4).

III. Arm lymphedema at 1 year as measured by arm circumference. IV. Arm range of motion at 1 year as measured by goniometry. V. Quality of life at 1 year as measured by FACT-B+4. VI. Percent increase in arm strength as measured by one repetition maximum at 1 year.

VII. Change in weight and body mass index (BMI) 1 year after completion of radiation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive usual care for 6 weeks during radiation therapy and for 12 weeks after completion of radiation therapy.

ARM II: Patients undergo a supervised aerobic and strength training exercise session over 40-60 minutes 3 times weekly for 6 weeks during radiation therapy and for 12 weeks after completion of radiation therapy.

After completion of study, patients are followed up at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-III breast cancer
* Prior surgery including lumpectomy or mastectomy and sentinel node biopsy or axillary lymph node dissection
* Prior chemotherapy in the neoadjuvant or adjuvant setting
* Radiation plan consisting of regional nodal radiation
* Must be suitable for an exercise program

Exclusion Criteria:

* Serious underlying medical comorbidity such as uncontrolled hypertension, cardiovascular disease, pulmonary disease, psychiatric illness, or any other condition for which the patient is not approved for exercise by their physician
* Physical handicap that would prevent participation in program
* Patients with metastatic breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete 70% of all exercise sessions throughout the supervised program during and after radiation therapy (Pilot) | Up to 1 year
  determine the feasibility of conducting an exercise program during and after radiation therapy and to determine what percent of patients will complete the exercise program.
Percent increase in fitness as measured by the 6 minute walk test in patients randomized to exercise program (Phase II) | At 1 year
  Will be compared to usual care group.

SECONDARY OUTCOMES:
Arm lymphedema as measured by arm circumference | Baseline up to 1 year
  Lymphedema will be classified into 3 stages. Stage I edema is reversible and characterized by pitting edema, increase in arm girth, and heaviness. Stage II is characterized by a spongy consistency of the arm without pitting edema. Stage III is the most advanced stage, lymphostatic elephantiasis
Arm range of motion as measured by goniometry | Baseline up to 1 year
  Shoulder flexion, external and internal rotation, and abduction will be measured.
Change in weight and BMI | Baseline up to 1 year
  BMI will be measured to evaluate body composition using the metric formula weight (kg)/ height 2 (m2).
Percent adherence to exercise as measured by the International Physical Activity Questionnaire and exercise logs | Baseline up to 1 year
  Duration of exercise will be calculated based on questionnaire and exercise log. Percentage of exercise adherence at 1-year follow-up will be compared between two groups. Generalized linear models will be utilized to model follow-up as a function of baseline and group.
Percent increase in arm strength as measured by one repetition maximum | Baseline up to 1 year
  Change in strength from baseline to post-intervention and follow-up will be obtained.
Quality of life as measured by FACT-B+4 | Baseline up to 1 year
  The FACT B + 4 has been shown to have good internal consistency and stability. It is a 40 item Likert scale questionnaire with subscales (0 - 4) for physical well being, social/family well being, emotional well being, function well being, and 4 specific questions related to arm symptoms.
Subjective arm health as measured by FACT-B+4 | Baseline up to 1 year
  The FACT B + 4 has been shown to have good internal consistency and stability. It is a 40 item Likert scale questionnaire with subscales (0 - 4) for physical well being, social/family well being, emotional well being, function well being, and 4 specific questions related to arm symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Beyer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu